CLINICAL TRIAL: NCT01742234
Title: Renal and Lung Living Donors Evaluation (RELIVE) Informed Consent Study
Brief Title: RELIVE Informed Consent Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT RELIVE 03
Record Dates: First submitted 2012-11-28; First posted 2012-12-05 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Living Donors; Tissue Donors
MeSH Terms: interventions — Tissue and Organ Procurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Kidney Donors: People who will donate a kidney at the University of Minnesota, Mayo Clinic, or University of Alabama
  Interventions: Procedure: Organ Donation
- Lung Donors: People who will donate a lung at the Washington University School of Medicine or the University of Southern California
  Interventions: Procedure: Organ Donation

INTERVENTIONS:
Procedure: Organ Donation — People in this study will donate either a lung or kidney

SUMMARY:
An organ transplant is frequently the best option and, in some cases, the only option to save the lives of transplant recipients. Receiving an organ from a living donor eliminates the need to wait for a deceased donor, an option that many transplant recipients do not survive. However, donating an organ presents health concerns to the donor as well. This study will use surveys to evaluate the understanding of risk and psychological pressure that living organ donors felt when making the decision to donate. It will also compare participants' answers across geographic, racial and socio-economic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Living donor of a kidney or lung

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who will be donating at kidney at the University of Minnesota, Mayo Clinic, or University of Alabama or people who will be donating a lung at University of Washington Medical School or the University of Southern California
Sampling Method: Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Questionnaire Score 1 | Change from 1 week prior to donation and 3 months after donation
  Feelings of pressure to donate an organ on a 4-point scale e.g.; "1: No pressure" to "4: A lot of pressure."
Questionnaire Score 2 | Change from 1 week prior to donation and 3 months after donation
  Understanding of the donor screening process on a 4-point scale e.g.; "1: No understanding" to "4: Full understanding."
Questionnaire Score 3 | Change from 1 week prior to donation and 3 months after donation
  Understanding of medical and psychosocial consequences of organ donation on a 4-point scale e.g.; "1: No understanding" to "4: Full understanding."

SECONDARY OUTCOMES:
Questionnaire Score Secondary Endpoint 1 | Change from 1 week prior to donation and 3 months after donation
  Understanding of short-term medical risks of donation answered on a 4-point scale e.g.; "1: No understanding" to "4: Full understanding."
Questionnaire Score Secondary Endpoint 2 | Change from 1 week prior to donation and 3 months after donation
  Understanding of long-term medical risks of donation expressed by donors on a scale of 1 to 4 e.g.; "1: No understanding" to "4: Full understanding."
Questionnaire Score Secondary Endpoint 3 | Change from 1 week prior to donation and 3 months after donation
  Understanding of psychological risks of donation expressed by donors on a scale of 1 to 4 e.g.; "1: No understanding" to "4: Full understanding."
Questionnaire Score Secondary Endpoint 4 | Change from 1 week prior to donation and 3 months after donation
  Understanding that recipients may have variable outcomes as expressed by donors on a scale of 1 to 4 e.g.; "1: No understanding" to "4: Full understanding."

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Valapour, MD, Study Chair — University of Minnesota, Center for Bioethics

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Valapour M, Kahn JP, Bailey RF, Matas AJ. Assessing elements of informed consent among living donors. Clin Transplant. 2011 Mar-Apr;25(2):185-90. doi: 10.1111/j.1399-0012.2010.01374.x. Epub 2010 Dec 16. PMID 21158924
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY292 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY292 — ImmPort study identifier is SDY292
- Available data/document: Study Protocol: SDY292 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY292 — ImmPort study identifier is SDY292. The study protocol is available in the Design tab section.